CLINICAL TRIAL: NCT02085525
Title: A Randomized Comparative Study of a Weekly Versus Every Other Week Nurse Practitioner-led Symptom Management Clinic for Head and Neck Cancer Patients Undergoing Concurrent Chemotherapy and Radiation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2014.018; HUM00085186 (Other: University of Michigan)
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weekly NP Visits (Other): 100 HNC (Head and Neck Cancer) patients seen weekly in a Nurse Practitioner (NP) led symptom management clinic for supportive care.
  Interventions: Other: Nurse Practitioner Clinic
- Every Other Week NP Visits (Other): 100 HNC (Head and Neck Cancer) patients seen every other week in a Nurse Practitioner (NP) led symptom management clinic for supportive care.
  Interventions: Other: Nurse Practitioner Clinic

INTERVENTIONS:
Other: Nurse Practitioner Clinic — The nurse practitioner (NP) clinic is staffed by two NPs, one registered nurse, and several medical assistants. Patients can be seen by either NP during their treatment course. Patients will be scheduled to be seen in the (NP) clinic based on randomization assignment.
  Each clinic visit focuses on specific concerns and toxicities of the patient and their significant other. This will include physical as well as psychological, social and spiritual needs.

SUMMARY:
A retrospective chart review of patients receiving concurrent chemoradiotherapy for oropharynx cancer was performed to compare clinical data for patients treated prior to the initiation of the NP clinic with those subsequently seen weekly in the NP clinic. The variables studied included; rate of hospitalization, dose completion and dose reductions. The results revealed an overall improvement in all variables for those patients seen in the weekly NP clinic.

To further analyze this data a randomized, prospective study is proposed to validate the findings of the retrospective study. It is predicted that a weekly NP led clinic will decrease costly hospitalizations, increase patient treatment completion and improve overall patient quality of life and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of stage III or IV HNC
* Are initiating concurrent chemotherapy and radiation
* Are able and willing to sign informed consent
* Ages 18 years or older
* ECOG (Eastern Cooperative Oncology Group) score of 0 or 1 (The ECOG score attempt to quantify cancer patients' general well-being and activities of daily life)
* Able to read and complete the required survey

Exclusion Criteria:

* Cannot provided informed consent
* Any medical or psychiatric illness which in the opinion of the principal investigator would compromise the patient's ability to tolerate this treatment.
* Have a history of prior cancer within past 5 years (excluding non-melanoma skin cancer)
* Are unwilling or unable to complete the required QOL (Quality of Life) survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients that Experience a "Problem" during Cancer Treatment | 11 weeks
  A "problem" includes any one of three events: dose reduction, inability to complete treatment, or toxicity related hospitalization. Patients are assigned a 1 if any of these events occurs at least once during treatment or are assigned 0 if they complete treatment with no dose reductions or toxicity related hospitalizations. When data is analyzed and reported, the problem rate will be summarized along with the each individual negative component.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Worden, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States